CLINICAL TRIAL: NCT06106178
Title: A Novel Serious Game as an Alternative for Teaching Basic Point-of-Care Transthoracic Echocardiography Skills
Acronym: SLOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Josef Michael Lintschinger, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1289/2023
Record Dates: First submitted 2023-04-03; First posted 2023-10-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-05

CONDITIONS: Echocardiography; Education, Medical
Keywords: Echocardiography; Education, Medical; Anesthesiology; Critical Care

STUDY DESIGN:
Intervention Model Description: Participants will attend a 90-minute workshop to learn the basics of point-of-care echocardiography. They will then be required to perform standardized transthoracic echocardiography before and after a two-week training period, which will be scored by blinded experts. During the training phase, one group will practice the hand-eye coordination required for echocardiography using an ultrasound simulator, while the second group will practice the same content using a serious video game. In addition, questionnaires will be used to collect additional data from the participants.
Who Masked: Outcomes Assessor
Masking Description: The POCUS examinations are videotaped without the possibility of identifying the participant. A camera visually records the movements of the ultrasound probe and the participant's hand, while a pen is used to mark the appropriate structures on the frozen ultrasound images. The audio recordings of these videos are transcribed and presented to the evaluators in written form only. After all participants have completed the baseline assessment, these two videos from each participant will be edited together and can be presented to the experts for evaluation as a compact video along with the transcribed audio recordings. In addition, the videos and audio transcripts presented to the experts will be labeled with randomly generated numbers for scoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simulator for Basic Ultrasound Skills (Other): Basic course of a traditional ultrasound simulator focusing on hand-eye coordination
  Interventions: Other: Simulator for Basic Ultrasound Skills
- Serious Video Game (Other): Serious video game "Underwater" that focuses on hand-eye coordination training using a 3D-printed ultrasound probe for maneuvering.
  Interventions: Other: Serious Video Game

INTERVENTIONS:
Other: Simulator for Basic Ultrasound Skills — Basic course of a traditional ultrasound simulator focusing on hand-eye coordination
  Arms: Simulator for Basic Ultrasound Skills
Other: Serious Video Game — The serious video game "Underwater" uses a 3D-printed ultrasound probe for maneuvering. During gameplay, coins must be collected in an underwater world using the aforementioned simulated ultrasound probe. The main focus of this game is to improve hand-eye coordination while using an ultrasound probe.
  Arms: Serious Video Game

SUMMARY:
The goal of this clinical trial is to compare different digital learning methods for teaching basic skills in point-of-care transthoracic echocardiography to medical students.

The main question it aims to answer is:

• Is a novel digital learning tool, such as a serious video game, non-inferior to traditional ultrasound simulator teaching methods in the context of basic point-of-care transthoracic echocardiography skills training?

Participants will train basic point-of-care ultrasound skills using either a traditional basic ultrasound simulator course or the serious video game "Underwater". Both methods focus on training hand-eye coordination, which is particularly important in transthoracic echocardiography. To compare the performance of the participants, a baseline assessment will be performed before and a final assessment after the two-week training period.

DETAILED DESCRIPTION:
Point-of-care ultrasound education follows non-standardized teaching and learning methods. In many cases, ultrasound is practiced directly on patients without proper training, or ultrasound simulators are used. However, these simulators are expensive to purchase and are not always readily available to students. In addition, there are a growing number of new digital tools, such as serious video games, that aim to deliver the same content in a more accessible and cost-effective manner. However, in the field of point-of-care echocardiography, there is still little scientific evidence to support their use.

This single-blind, prospective, randomized, controlled, non-inferiority trial aims to demonstrate the non-inferiority of a serious video game compared to conventional simulator-based training of basic echocardiography skills to make ultrasound training more accessible to every trainee.

Only medical students who already have the necessary anatomical knowledge but no experience with ultrasound diagnostics will be recruited to participate in this study. Participants will attend a 90-minute workshop to learn the basics of point-of-care echocardiography. They will then be required to perform standardized transthoracic echocardiography before and after a two-week training period, which will be scored by blinded experts. During the training phase, one group will practice the hand-eye coordination required for echocardiography using an ultrasound simulator, while the second group will practice the same content using a serious video game. In addition, questionnaires will be used to collect additional data from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Medical student at the Medical University of Vienna (Medicine Degree Program)
* ≥18 years
* Basic knowledge of anatomy (completed Block 2 of the MUV curriculum)

Exclusion Criteria:

* Previous experience using an ultrasound device

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will be asked about their gender identity and will be randomized equally per gender to the control or intervention group.
Enrollment: 120 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in the participants' modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment | Two-week change from baseline to final assessment score
  The primary outcome measure is the difference in the participant's modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the participants' baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.

SECONDARY OUTCOMES:
Gender differences in modified Objective Structured Assessment of Ultrasound Skill (OSAUS) scores between the baseline and final assessment | evaluation within 3 weeks after study completion
  A two-factorial analysis of variance model (including an interaction term) will be used to determine the influence of gender in the difference of the modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. To adjust for potential imbalances between the randomized groups, the HEXACO (a measure of the six major dimensions of personality; H: Honesty-Humility; E: Emotionality; X: eXtraversion; A: Agreeableness (versus Anger); C: Conscientiousness; O: Openness to Experience) subscale of openness to experience (ranging from 1 to 5, with higher scores indicating more openness to experience) and the Technology Readiness Score (ranging from 1 to 5, with higher scores indicating more technology readiness) were included as covariates in the ANCOVA model.
Group effects on gender differences in modified Objective Structured Assessment of Ultrasound Skill (OSAUS) scores | evaluation within 3 weeks after study completion
  A two-factorial analysis of variance model (including an interaction term) will be used to determine the potential modifying effect of gender on the training effect, which is calculated as the difference in the participant's total modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the participant's baseline assessment and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. To adjust for potential imbalances between the randomized groups, a scale for openness to experience (ranging from 1 to 5, with higher scores indicating more openness to experience) and the Technology Readiness Score (ranging from 1 to 5, with higher scores indicating more technology readiness) are included as covariates in the ANCOVA model.
Time to complete the baseline assessment | up to 10 minutes
  The maximum time (minutes and seconds) to complete the baseline assessment is set to 10 minutes. Therefore, times between 0 and 10 minutes can be measured.
Time to complete the final assessment | up to 10 minutes
  The maximum time (minutes and seconds) to complete the final assessment is set to 10 minutes. Therefore, times between 0 and 10 minutes can be measured.
Spearman correlation coefficients between the time taken and the participants learning progress | evaluation within 3 weeks after study completion
  Spearman correlation coefficients between the time taken for the final assessment and the difference in the participant's modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the participant's baseline final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.
Group difference in modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score points for each objective | Two-week change from baseline to final assessment score
  Possible scores range from 1 to 4 points per objecitve, with higher scores indicating better performance.
  Objectives are: applied knowledge of ultrasound equipment; image optimization; systematic examination; interpretation of images
Subjective confidence of participants in the use of point-of-care ultrasound (POCUS) in the context of transthoracic echocardiography after the training period | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating greater confidence
  (1: not confident; 2: rather not confident; 3: neither confident nor not confident; 4: confident; 5: very confident)
Group difference in cognitive load while performing the final assessment as opposed to the respective cognitive load at the baseline assessment | Two-week change from baseline to final assessment
  Global National Aeronautics and Space Administration (NASA) Task-Load-Index ranging from 0 to 100. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective score of the final assessment is calculated. Higher scores are indicating higher cognitive load.
Group difference in cognitive load (per objective) while performing the final assessment as opposed to the respective cognitive load at the baseline assessment | Two-week change from baseline to final assessment
  National Aeronautics and Space Administration (NASA) Task-Load-Index per objective, ranging from 0 to 100. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective score of the final assessment is calculated.
  Objectives are: (mental demand, physical demand, temporal demand, performance, effort, frustration). Higher scores are indicating higher mental demand/higher physical demand/ higher temporal demand/worse performance/more effort/more frustration).
Subjective desire for for more new digital tools in medical education before and after the training period | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating more desire
  (1: no desire; 2: rather not a desire; 3: neither a desire nor not a desire; 4: a desire; 5: a strong desire)
Frequency of playing video games for fun in the past 12 months before the study | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating higher frequency
  (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily)
Frequency of playing video games for educational purposes in the past 12 months before the study | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating higher frequency
  (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily)
Frequency of playing video games for fun between the ages of 6 and 18 | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating higher frequency
  (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily)
Frequency of playing video games for educational purposes between the ages of 6 and 18 | evaluation within 3 weeks after study completion
  5-point Likert Scale, with higher scores indicating higher frequency
  (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily)
Correlation between the frequency of playing video games for fun in the past 12 months before the study and the learning progress | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the difference in the participants' modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.
Correlation between the frequency of playing video games for educational purposes in the past 12 months before the study and the difference in the learning progress | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the difference in the participants' modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.
Correlation between the frequency of playing video games for fun between the ages of 6 and 18 and the difference in the learning progress | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the difference in the participants' modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.
Correlation between the frequency of playing video games for educational purposes between the ages of 6 and 18 and the difference in the learning progress | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the difference in the participants' modified Objective Structured Assessment of Ultrasound Skill (OSAUS) score between the baseline and final assessment. Possible assessment scores range from 4 to 20 points, with higher scores indicating better performance. Each participant's baseline assessment score is his or her individual baseline score, from which the difference to the respective final assessment score is calculated.
Correlation between the frequency of playing video games for fun in the past 12 months before the study and the desire for more digital tools in medical education before and after the training period within the study | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the desire for more digital tools in medical education before and after the training period of this study. This desire will be measured with a 5-point Likert Scale, with higher scores indicating more desire (1: no desire; 2: rather not a desire; 3: neither a desire nor a desire; 4: a desire; 5: a strong desire)
Correlation between the frequency of playing video games for educational purposes in the past 12 months before the study and the desire for more digital tools in medical education before and after the training period within the study | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the desire for more digital tools in medical education before and after the training period of this study. This desire will be measured with a 5-point Likert Scale, with higher scores indicating more desire (1: no desire; 2: rather not a desire; 3: neither a desire nor a desire; 4: a desire; 5: a strong desire)
Correlation between the frequency of playing video games for fun between the ages of 6 and 18 and the desire for more digital tools in medical education before and after the training period within the study. | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the desire for more digital tools in medical education before and after the training period of this study. This desire will be measured with a 5-point Likert Scale, with higher scores indicating more desire (1: no desire; 2: rather not a desire; 3: neither a desire nor a desire; 4: a desire; 5: a strong desire)
Correlation between the frequency of playing video games for educational purposes between the ages of 6 and 18 and the desire for more digital tools in medical education before and after the training period within the study. | evaluation within 3 weeks after study completion
  Spearman correlation between the frequency of playing video games, measured with a 5-point Likert Scale, with higher scores indicating higher frequency (1: never; 2: less than once a week; 3: once a week; 4: more than once a week; 5: daily) and the desire for more digital tools in medical education before and after the training period of this study. This desire will be measured with a 5-point Likert Scale, with higher scores indicating more desire (1: no desire; 2: rather not a desire; 3: neither a desire nor a desire; 4: a desire; 5: a strong desire)
Subjective feeling of learning progress during the training period | evaluation within 3 weeks after study completion
  5-point Likert Scale measuring the subjective feeling of learning progress with the digital training tool within the randomized group
  (1: not helpful; 2: rather not helpful; 3: neither helpful nor not helpful; 4: rather helpful; very helpful)
Subjective level of frustration during the training period | evaluation within 3 weeks after study completion
  5-point Likert Scale measuring the subjective feeling of frustration while using the digital training tool within the randomized group
  (1: no frustration; 2: rather not frustrated; 3: neither frustrated nor not frustrated; 4: rather frustrated; 5: very frustrated)
Subjective level of enjoyment during the training period | evaluation within 3 weeks after study completion
  5-point Likert Scale measuring the subjective feeling of frustration while using the digital training tool within the randomized group
  (1: no enjoyment; 2: rather no enjoyment; 3: neither enjoyment nor no enjoyment; 4: rather an enjoyment; 5: strong enjoyment)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Serious Video Game "Underwater" — https://www.sfinxgames.com/projectPages/projectpage_underwater.shtml